CLINICAL TRIAL: NCT02546804
Title: Evaluate the Efficacy of Potassium Permanganate Mouthwash and Hot Salt Water Mouthwash and Their Comparison With Chlorhexidine Mouthwash on Plaque Index,Gingival Index and Periodontal Probing Depth
Brief Title: A Clinical Trial to Study the Effects of Two Home Made Mouthwashes in Patients With Gum Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Agrima Singh, P.G. Student, Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCDIndore
Record Dates: First submitted 2015-08-26; First posted 2015-09-11 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis | interventions — Potassium Permanganate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HOT SALT WATER (Experimental): 3% HOT SALT WATER , 25ml used for rinsing for 60 sec, twice daily for 60 days.
  Interventions: Procedure: HOT SALT WATER
- POTASSIUM PERMANGANATE (Experimental): 0.01% POTASSIUM PERMANGANATE, 10ml used for rinsing for 60 sec, twice daily for 60 days.
  Interventions: Procedure: POTASSIUM PERMANGANATE
- CHLORHEXIDINE (Active Comparator): 0.2% CHLORHEXIDINE, 10ml used for rinsing for 60 sec, twice daily for 60 days.
  Interventions: Procedure: CHLORHEXIDINE

INTERVENTIONS:
Procedure: HOT SALT WATER — 25ml mouthwash will be rinsed for 60sec), twice daily for 60 days The subjects then will be recalled for measuring the data's after 2weeks, 4weeks, 6weeks and 8weeks.
  Arms: HOT SALT WATER
Procedure: POTASSIUM PERMANGANATE — 10ml mouthwash will be rinsed for 60sec), twice daily for 60 days The subjects then will be recalled for measuring the data's after 2weeks, 4weeks, 6weeks and 8weeks.
  Arms: POTASSIUM PERMANGANATE
Procedure: CHLORHEXIDINE — 10ml mouthwash will be rinsed for 60sec), twice daily for 60 days The subjects then will be recalled for measuring the data's after 2weeks, 4weeks, 6weeks and 8weeks.
  Arms: CHLORHEXIDINE

SUMMARY:
Periodontal Disease is a ubiquitous in nature affecting about 80% population of India. The Periodontal Disease is a multifactorial but the dental plaque is considered as main etiological agent.The dental plaque, a adhesive bacterial coating accumulate around and in between teeth, if not removed by effective daily brushing and flossing, plaque can cause Gum infection and tooth loss. Though, many scientific periodontal procedures are available to get the treatment but because of lack of man power and poor socioeconomic condition it is not possible for every group of population in our India.

DETAILED DESCRIPTION:
The need exist for continued research to find the use of home made mouthwashes in preventing periodontal diseases. Although, Chlorhexidine mouthwash is regarded as Gold standard mouthwash as antiplaque but have some limitations like cost factor and side effects like staining of teeth, loss of taste, oral mucosal ulcerations,paresthesia and may enhanced supragingival calculus formation. Use of various indigenous products and home made preparations are easily available and are being used since ancient time in India and still in practice in various parts of India especially rural and remote areas.

At the same time the use of potassium permanganate is still in practice in various parts of India and also it was in practice before the availability of Chlorhexidine, povidone iodine and other antiseptic solutions, as they are used since about 30 years only. Use of hot salt water rinsing is in practice especially to reduce the symptoms of various throat infections such as pharyngitis, tonsillitis and also to improve oral hygiene.It is also being used in oral surgery and their effects are also mention in literature.

Hence, the aim of this study is to assess and compare the efficacy of home made remedies like hot salt water and potassium permanganate as a mouthwash in reducing Plaque accumulation and improving Gingival conditions with Gold standard Chlorhexidine mouthwash if found effective may be used as affordable mouthwash for the benefit of population of India.

ELIGIBILITY:
Inclusion Criteria:

* Subject of Chronic Generalized Gingivitis and Mild Generalized Periodontitis.
* Not undergone any major periodontal treatment earlier in last 06 months .
* Otherwise Clinically Healthy Patient.

Exclusion Criteria:

* Subjects with significant systemic diseases (e.g. Diabetes Mellitus, Cancer or Coronary heart disease etc.).
* Pregnant or lactating women.
* Smoker.
* Patients on anti-inflammatory drugs or antibiotics
* Patients allergic to any material used for the study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plaque Index | baseline
  4 sites of all tooth is observed

SECONDARY OUTCOMES:
Plaque Index | 2weeks
  4 sites of all tooth is observed
Plaque Index | 4weeks
  4 sites of all tooth is observed
Plaque Index | 6weeks
  4 sites of all tooth is observed
Plaque Index | 8weeks
  4 sites of all tooth is observed
Gingival Index | baseline
  4 sites of all tooth is observed
Gingival Index | 2weeks
  4 sites of all tooth is observed
Gingival Index | 4weeks
  4 sites of all tooth is observed
Gingival Index | 6weeks
  4 sites of all tooth is observed
Gingival Index | 8weeks
  4 sites of all tooth is observed
Periodontal Probing Depth | baseline
  6 sites of all tooth is observed
Periodontal Probing Depth | 2weeks
  6 sites of all tooth is observed
Periodontal Probing Depth | 4weeks
  6 sites of all tooth is observed
Periodontal Probing Depth | 6weeks
  6 sites of all tooth is observed
Periodontal Probing Depth | 8weeks
  6 sites of all tooth is observed

CONTACTS AND LOCATIONS:
Overall Officials: agrima singh, Principal Investigator — Government College of Dentistry
Locations (1):
- Agrima Singh, Indore, Madhya Pradesh, India

REFERENCES:
- [Background] Resende MM, Rocha CA, Correa NF, Veiga RR, Passos SJ, Novo NF, Juliano Y, Damasceno CA. Tap water versus sterile saline solution in the colonisation of skin wounds. Int Wound J. 2016 Aug;13(4):526-30. doi: 10.1111/iwj.12470. Epub 2015 Jun 8. PMID 26059709
- [Background] Supranoto SC, Slot DE, Addy M, Van der Weijden GA. The effect of chlorhexidine dentifrice or gel versus chlorhexidine mouthwash on plaque, gingivitis, bleeding and tooth discoloration: a systematic review. Int J Dent Hyg. 2015 May;13(2):83-92. doi: 10.1111/idh.12078. Epub 2014 Jul 24. PMID 25059640